CLINICAL TRIAL: NCT05634109
Title: Whole Blood vs. Blood Components Therapy in the Hemostatic Resuscitation of Severe Trauma Patients: An Open-label, Randomized, Controlled Clinical Trial
Brief Title: Whole Blood in Trauma Patients With Hemorrhagic Shock
Acronym: WEBSTER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: University of Pittsburgh (Other); Hospital Universitario del Valle Evaristo Garcia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1938
Record Dates: First submitted 2022-11-16; First posted 2022-12-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Trauma; Trauma Injury; Trauma, Multiple
Keywords: whole blood; Blood Transfusion; Blood Component Transfusion; Hemorrhage; Advanced Trauma Life Support Care; Hemostatic resuscitation
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries; Multiple Trauma; Hemorrhage | interventions — Blood Transfusion

STUDY DESIGN:
Intervention Model Description: Single center, Controlled, Randomized, and Open label therapeutic trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Blood (Experimental): Leukoreduced whole blood with a platelet-sparing filter. Participants will be transfused with 3 whole blood units. If the participant requires, an additional transfusion pack composite by 3 whole blood units will be administered.
  Interventions: Biological: Transfusion of blood products
- Blood Components Therapy (Active Comparator): 1:1:1 ratio of red blood cells unit, plasma unit, and platelets unit. Participants will be transfused with 3 red blood cell units, 3 fresh frozen plasma units, and 3 platelets units. A second intervention with the same ratio can be transfused to participants if they require it.
  Interventions: Biological: Transfusion of blood products

INTERVENTIONS:
Biological: Transfusion of blood products — The intervention will be either a) administration of 6 units of whole blood or b) administration of blood component therapy in the proportion of 6:6:6 units of red blood cells, plasma, and platelets.

SUMMARY:
This study aims to evaluate among trauma patients with hemorrhagic shock the clinical impact of hemostatic resuscitation between whole blood vs. blood components therapy in the following outcomes in a hierarchical analysis: mortality at 28 days and evolution of organ dysfunction.

DETAILED DESCRIPTION:
Background: Hemostatic resuscitation is a mainstay in the management of trauma patients. Factors such as blood loss and tissue injury contribute to coagulation and hemodynamic status imbalances. Hemorrhage remains a leading cause of death in trauma patients, despite advances in strategies such as damage control surgery, massive transfusion protocol, and intensive care.

Conventional therapy for hemostatic resuscitation is a blood transfusion seeking a 1:1:1 ratio of red blood cells, plasma, and platelets. However, this ratio has disadvantages in clinical practice, especially in low-resource settings. Whole blood transfusion can contribute to maintaining a physiological rate of cells, clotting factors, and hemostatic properties. Advances in the whole blood elucidated a new opportunity for its implementation in civilian trauma centers. However, the effect of initial resuscitation with whole blood in trauma patients is unclear. This study aims to determine the effect of hemostatic resuscitation using whole blood on mortality and evolution of organ dysfunction in severe trauma patients compared to blood components therapy. This clinical trial attempts to resolve the debate and uncertainty of using whole blood vs. blood components.

Study Design: An open-label, randomized, prospective, single-center and controlled trial will be performed. This study will be included prospectively randomized severe trauma patients who require a blood transfusion. Randomization can assign participants to the experimental arm, transfusing them with 3 units of whole blood. If the participant continues requiring transfusions, the second intervention of 3 units of whole blood can be administered. On the contrary, the randomization can assign to the control arm, where the participant will receive 3 red blood cell units, 3 fresh frozen plasma units, and half of a platelets apheresis, equivalent to 3 platelets units. If required, a second intervention with the same ratio can be transfused to participants.

The primary outcome is a hierarchical composite outcome based on mortality at 28 days and the evolution of organ dysfunction. Organ dysfunction will be measured as the difference in the score between the fifth and first days of the SOFA (Sequential Organ Failure Assessment). Secondary outcomes are mortality, coagulopathy profile, intensive care unit free days, length of hospital stay free days, and volumes of transfusion requirements. Safety outcomes are complications related to transfusion (anaphylaxis, acute hemolytic reaction, acute lung injury) and complications related to trauma patients (acute distress respiratory syndrome, pulmonary embolism, deep vein thrombosis, acute kidney injury with or without dialysis, stroke, myocardial infarction, cardiac arrest, sepsis, abdominal complications, abdominal compartment syndrome)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* Activating institutional trauma code for trauma patients with hemorrhagic shock.
* Candidate for massive transfusion (Patient with an Assessment Blood Consumption (ABC) Score ≥ 2 or at the discretion of the treating physician)
* Concurrent availability of whole blood or blood component therapy

Exclusion Criteria:

* More than 4 hours from trauma to hospital admission
* More than 2 hours from hospital admission to randomization
* Transfusion of more than one packed red blood cell unit prior to randomization.
* Patients who have undergone surgery (laparotomy, thoracotomy, or sternotomy) before hospital admission.
* In-extremis patients with devastating injuries (expected to die within 60 minutes).
* Blood group other than to O or A and positive Rh factor
* Severe traumatic brain injury in which neurosurgical intervention is futile (partial decapitation, massive intracranial hemorrhage, or transcranial gunshot wounds).
* Burns over 20% of the total body surface area.
* Suspected airway burn.
* Cardiopulmonary resuscitation (CPR) before arrival at the ED.
* CPR for more than 5 minutes before randomization.
* Do not resuscitate order.
* Incarcerated/prisoners.
* Known pregnancy in the ED.
* Patient or legal representative who refuse to participate in clinical research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is a hierarchical outcome consisting of mortality at 28 days post-randomization and evolution of organ dysfunction (difference of Sequential Organ Failure Assessment (SOFA) score between day 1 and day 5 post-randomization). | 28 days post ED admission
  The primary outcome is a hierarchical composite outcome that will be analyzed using the Win-Ratio test. The first level will be 28-day mortality. The "winner" will be the participant who survival; in case of a tie, the second level will be the difference in SOFA score between fifth and first day. The "winner" will be participant with the lowest difference.

SECONDARY OUTCOMES:
24-hour mortality | First 24 hours post ED admission.
  The occurrence of deaths in the first 24 hours post-ED admission and we will document and record the time of death in hours.
In-hospital mortality | 28 days post ED admission
  The occurrence of deaths during the hospital stays post-ED admission, and we will document and record the time of death in days.
Multiple organ dysfunction incidence | 1-day / 3-day / 5-day / 7-day post-ED admission
  Multiple organ dysfunction is a score ≥ 3 in two or more systems evaluated by SOFA score.
Evolution of Coagulopathy | Admission - 3 hours - 6 hours - 24 hours post-ED admission
  We will evaluate the values of INR, fibrinogen, and MA-TEG during the admission and the first 24 hours post-ED admission.
Intensive care unit-free days | 28-days post-ED admission
  ICU-free days
Hospital length stay-free days | 28-days post-ED admission
  Hospital length stay-free days
Blood transfusion requirements during the first 24 hours | Time frame 3 hours / 6 hours / 12 hours / 24 hours
  The number of units of whole blood or blood components transfused. Comparisons will be according to the following references:
  * 1 Unit of Whole blood = 1 Unit of packed red blood cells.
  * 1 Unit of Whole Blood = 1 Unit of Plasma
  * 1 Unit of Whole Blood = 1 Unit of Platelets
Proportion of participants with transfusional adverse reactions | 28-days post-ED admission
  We will document transfusional adverse reactions such as acute hemolytic reaction, anaphylaxis, non-hemolytic febrile transfusion reaction, allergy, and potassium and calcium electrolyte disorders.
Proportion of participants with adverse reactions | 28-days post-ED admission
  We will document adverse reactions such as acute lung injury, acute respiratory distress syndrome, pulmonary embolism, deep vein thrombosis, acute kidney injury with or without dialysis, stroke, myocardial infarction, cardiac arrest, sepsis, abdominal complications, and abdominal compartment syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Alberto F Garcia, MD MSc, Principal Investigator — Fundacion Clinica Valle del Lili; Carlos A Ordoñez, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Clinica Valle del Lili, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Derived] Garcia AF, Caicedo Y, Gempeler A, Vallecilla L, Macia C, Orlas C, Fernandez MI, Lancheros-Ramirez P, Quintero M, Hernandez E, Vargas S, Cardenas-Perez L, Ariza F, Zarama V, Carvajal S, Billefals E, Sanchez A, Badiel M, Rosso F, Granados M, Albornoz LA, Puyana JC, Ospina-Tascon G, Ordonez CA. Transfusion of modified whole blood versus blood components therapy in patients with severe trauma: Randomized controlled trial protocol (WEBSTER trial). Injury. 2025 May;56(5):112173. doi: 10.1016/j.injury.2025.112173. Epub 2025 Jan 23. PMID 40087111